CLINICAL TRIAL: NCT06509555
Title: Establishment of Serum TK1 Combined With MRI to Predict Pathological Remission of Breast Cancer With Neoadjuvant Chemotherapy
Brief Title: Correlation Between Serum TK1 and Pathological Remission of Breast Cancer With Neoadjuvant Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024.0716
Record Dates: First submitted 2024-07-13; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms; TK1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCR
  Interventions: Other: non-intervention
- non-PCR
  Interventions: Other: non-intervention

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
The levels and changes of sTK1 among different outcome groups in BCs with different molecular types were compared by stratification to explore whether sTK1 can be used as one of the tumor markers to predict pathological remission of NACT in BC patients.The changes of serum sTK1 level and ADC before surgery were continuously monitored, and combined with other clinicopathological factors, the pathological remission prediction model of NACT in BC patients was constructed and verified.

DETAILED DESCRIPTION:
Female patients diagnosed with breast cancer by breast biopsy and receiving neoadjuvant chemotherapy in our hospital from 2020 to 2024 were selected as the study objects, and their puncture pathology data, general clinical characteristics, hematology test data, imaging data and surgical pathology data were collected, and the data were collated for statistical analysis. The influencing factors of pCR after neoadjuvant therapy were determined by univariate and multivariate logistic regression analysis, and the nomogram and ROC curve were drawn. The model was verified internally through bootstrap resampling 1000 times, and the correction curve was drawn to evaluate the prediction ability of the model.

ELIGIBILITY:
Inclusion Criteria:

① The patient was diagnosed with breast cancer by biopsy, and there were complete pathological data. ② Complete the course of neoadjuvant chemotherapy; ③ After the end of neoadjuvant therapy, the operation was performed and the postoperative pathology was obtained; MRI and serum TK1 data were complete (baseline, after 2 cycles of chemotherapy, 4 cycles of chemotherapy, and 6 cycles of chemotherapy).

Exclusion Criteria:

① Distant metastasis at first diagnosis (stage IV); ② With other primary malignant tumors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient was diagnosed with breast cancer by biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Correlation analysis of serum TK1 and pathological remission of breast cancer with neoadjuvant chemotherapy | 2026.02

CONTACTS AND LOCATIONS:
Overall Officials: Qi Tang, doctor, Study Chair — Yunnan Cancer Hospital
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided